CLINICAL TRIAL: NCT00974246
Title: The Effect of Advair Diskus Treatment on Depression in Nursing Home Residents With COPD
Brief Title: The Effect on Depressive Symptoms in ECF Residents With COPD
Acronym: DISK-02
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Valley Medical Research (Other)
Responsible Party: Principal Investigator, Meenakshi Patel, MD, Meenakshi Patel, MD, Valley Medical Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DISK-02
Record Dates: First submitted 2009-09-08; First posted 2009-09-10 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Depression
Keywords: COPD; Depression; Nursing Home
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Depression | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD, ECF residents, Advair diskus (Experimental): open label treatment with Advair diskus in COPD patients
  Interventions: Drug: Advair diskus

INTERVENTIONS:
Drug: Advair diskus — Advair diskus 50/250 1 inhalation bid for 16 weeks

SUMMARY:
The purpose of this study is to assess the effect of treatment with Advair Diskus on depression using the Cornell depression scale in COPD patients in the nursing home.

DETAILED DESCRIPTION:
We are studying 35 residents in the ECF with a diagnosis of COPD. We are evaluating them for depressive symptoms using the Cornell Depression Scale and the MDS 3.0 section D. We are selecting patients who are not currently on treatment with Advair and starting them on Advair Diskus50/250 1 inhalation bid for a period of 16 weeks and reassessing the Cornell Depression SCale and MDS3.0 section D looking for any changes. We are also going to measure FEV1 and FVC using spirometry before treatment and at the end of 16 weeks. This is a pilot study. The numbers are not necessarily adequate to achieve statistical difference-we are looking for trends.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women nursing home residents up to age 95
* Stated diagnosis of COPD or FEV1/FVC <0.7 or being treated with an anticholinergic
* Presence of depressive symptoms as measured on MDS 3.0 Section D SUM
* Free from conditions likely to be fatal within six months
* Able to read or understand English
* Able and willing to provide informed consent or has a guardian/LAR who can provide informed consent

Exclusion Criteria:

* Currently pregnant
* Unable to read and understand English
* Free from conditions likely to be fatal within six months
* Enrolled in hospice
* New treatment with antidepressant within the last 90 days.
* Current or recent use (within the last 90 days) of Advair Diskus
* Unwilling or unable to provide informed consent
* Expected to be discharged within 3 months

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meenakshi Patel, MD, Principal Investigator — Valley Medical Research
Locations (2):
- United States (2):
  - Geriatric Medical Associates, Brooksville, Florida
  - Valley Medical Research, Centerville, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Population:: The study sample (n=27) were nursing home residents with either (1) a confirmed diagnosis of COPD, (2) an FEV1/FVC ratio <0.7 or (3) in treatment with anticholinergic drugs.
Period: Overall Study
Arm/Group | Study Population:
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Characteristics: Nursing Home residents with either a confirmed diagnosis of COPD or an FEV1/FVC ratio <0.7 or in treatment with anticholinergic drugs.
Arm/Group | Baseline Characteristics
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.7 (12.4)
Gender [Count of Participants; unit: Participants]
  Female | 20
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Effect of Treating COPD Patients With Advair Diskus for 16 Weeks on the Cornell Depression Scale or Section D SUM of the Minimum Data Set 3.0
Description: The Cornell Depression Scale ranges from 0-38, with a score 12 points or more indicating probable depression. Section D SUM o f the Minimum Date Set 3.0 is an assessment tool of health status for all residents (regardless of payer) of long-term care facilities certified to participate in Medicare or Medicaid. Scores range from 0 to 27, with a higher score indicating more depression.
Time Frame: 16 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Nursing Home Residents With COPD: The effect of Advair Diskus treatment on depression in nursing home residents with Chronic Obstructive Pulmonary Disease.
Arm/Group | Nursing Home Residents With COPD
Number analyzed (Participants) | 27
units on a scale
  Cornell Depression Scale | 8.7 [2 to 21]
  Section D SUM of the Minimum Data Set 3.0 | 10.8 [5 to 21]

2. Primary Outcome: To Determine if Changes in Pulmonary Function (FEC/FVC) Were Associated With a Reduction in Depression as Assessed by Using the Cornell Depression Scale or Section D SUM of the Minimum Data Set 3.0 During Advair Diskus Treatment.
Description: FEC is Forced Expiratory Capacity and FVC is Forced Vital Capacity. The Cornell Depression Scale ranges from 0-38, with a score 12 points or more indicating probable depression. Section D SUM o f the Minimum Date Set 3.0 is an assessment tool of health status for all residents (regardless of payer) of long-term care facilities certified to participate in Medicare or Medicaid. Scores range from 0 to 27, with a higher score indicating more depression.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nursing Home Residents With COPD
Number analyzed (Participants) | 27
units on a scale
  Cornell Depression Scale | 8.7 (5.0)
  Section D SUM of the Minimum Data Set | 10.8 (5.0)

3. Primary Outcome: Pulmonary Function FEC/FVC Ratio at 16 Weeks
Description: To measure whether pulmonary function, determined by the ratio between FEC (Forced Expiratory Capacity) and FVC (Forced Vital Capacity), improved during 16 weeks of Advair Diskus administration.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Study Population:
Number analyzed (Participants) | 27
ratio | 0.69 (0.13)

ADVERSE EVENTS:
Groups:
- Adverse Events: All enrolled subjects.
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=27)
Mental Status Change (Psychiatric disorders) | 1 (1) — Subject was sent to the Emergency Department for mental status changes. He was admitted for tests and observation. He was stabilized and discharged to the Nursing Home.
Increased Agitation with Combative Behaviors (Psychiatric disorders) | 1 (1) — Subject was sent to the Emergency Department for increased agitation with combative behaviors. She was admitted for observation and psychiatric treatment. She was stabilized and discharged to the Nursing Home.
Left Above the Knee Amputation (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject was sent to Emergency Department for possible Deep Vein Thrombosis (DVT). It was determined that she did have a DVT but it was too late to save the leg. An amputation was performed. Subject was stabilized & discharged to the Nursing Home.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=27)
Fall (Musculoskeletal and connective tissue disorders) | 11 (22)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 6 (6)
Bilateral Lower Extremity Edema (Blood and lymphatic system disorders) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruitis (Skin and subcutaneous tissue disorders) | 2 (2)
Right Hip Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Increased Aggression (Psychiatric disorders) | 2 (2)
Increased Restlessness (Psychiatric disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 7 (7)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 3 (3)
Cellulitis (Skin and subcutaneous tissue disorders) | 3 (3)
Headache (General disorders) | 2 (2)
Loose stool (Gastrointestinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypotension (Blood and lymphatic system disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Leg Pain (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No